CLINICAL TRIAL: NCT00202293
Title: Comparison of Combination Olanzapine and Lithium and Combination Chlorpromazine and Lithium in the Treatment of a First Manic Episode With Psychotic Features.
Brief Title: Comparison of Combination Olanzapine+Lithium or Chlorpromazine+Lithium in Treatment of First Manic Episode With Psychotic Features
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001.013
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2015-11

CONDITIONS: Bipolar Disorder; Schizoaffective Disorder
Keywords: Bipolar; Mania; Drug treatment; First episode; Psychosis; Therapy; Antipsychotic
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Mania | interventions — Olanzapine; Lithium; Chlorpromazine

ARMS (2):
- Lithium and olanzapine (Experimental)
  Interventions: Drug: Olanzapine; Drug: Lithium
- Lithium and chlorpormazine (Active Comparator)
  Interventions: Drug: Lithium; Drug: Chlorpromazine

INTERVENTIONS:
Drug: Olanzapine
  Arms: Lithium and olanzapine
Drug: Lithium
Drug: Chlorpromazine
  Arms: Lithium and chlorpormazine

SUMMARY:
Aim: In a population of first episode manic patients with psychotic features, we want to compare the side effect profile, the degree of adherence and the subjective well being, as well as the efficacy of two treatments: The standard treatment currently applied (lithium + chlorpromazine) and an alternative treatment more recently introduced (lithium + olanzapine). In addition, we want to study retrospectively the development of bipolar disorder and study prospectively the 6 and 12-month outcome of a cohort of patients presenting a first manic episode with psychotic features.

Research Background: While the efficacy of lithium in the treatment of acute mania has been established by numerous studies, it is also known that up to 50% of the patients fail to respond when it is prescribed alone. It is therefore common practice to complement the treatment, most commonly with antipsychotics and benzodiazepines. It has been suggested that antipsychotic agents are faster acting and are superior in controlling hyperactivity compared to lithium, whereas mood stabilisation is better achieved by lithium, Typical antipsychotics, such as chlorpromazine, may therefore be useful as adjunctive medication to mood stabilisers, especially within the first few weeks of treatment of acute mania, and for patients exhibiting psychotic symptoms or hyperactivity. They however can induce side effects (somnolence, dizziness, dry mouth, extrapyramidal side effects such as rigidity of the muscles, and possibly tardive dyskinesia (involuntary movements or contraction of muscles), as well as akathysia (sense of restlessness). They finally have been suspected to contribute to the occurrence of post-manic depression. Recent publications in chronic populations have shown that atypical antipsychotics, such as olanzapine, are also an effective adjunctive treatment. Olanzapine has the important advantage to induce a very low incidence of extrapyramidal side effects, including tardive dyskinesia. It can however induce somnolence, dizziness, dry mouth, and rather commonly weight gain. Moreover, some authors have reported that olanzapine might induce mania. Both treatments appear then to have positive effects as well as undesirable side effects. Our project is to compare them. The literature concerning first episode mania is sparse, particularly in the domain of pharmacotherapy. One retrospective study showed that 77% of the patients received antipsychotics at discharge and 25% at 6 months follow-up. No comparison has however been made between typical and atypical antipsychotics, and there are no specific treatment guidelines of first episode mania with psychotic features.

Project Summary: The hypothesis is that olanzapine and chlorpromazine will have a comparable efficacy as adjunctive treatment of the acute manic episode with psychotic features. We however think olanzapine will induce less side effects and will be better accepted by the patients, and therefore that the adherence to the treatment will be better than with chlorpromazine. We finally think the subjective sense of well being will be greater with olanzapine than with chlorpromazine.We will recruit 75 patients at the time of their first admission for mania with psychotic features at EPPIC. After signature of the informed consent, we will perform a baseline assessment first to confirm the diagnosis, and second to evaluate the level of psychopathology. The patients will then be randomly selected to receive either a treatment of lithium and olanzapine or a treatment of lithium and chlorpromazine. By the end of the study there will be 37 patients in each group.The patients will go through a baseline assessment including physical examination and usual laboratory investigation to exclude any physical illness. They will also go through a one-hour assessment of psychopathology. Between day 2 and 3 they will go through 2 hours of interview to reassess diagnosis and personal history. They will thereafter be assessed weekly for eight weeks on various dimensions: evolution of the intensity of the symptoms, appearance of depressive symptoms, occurrence of side effects and degree of adherence to the treatment, in an 1-hour interview. Subjective well being and quality of life will re evaluated at week 4 and 8, adding 45 minutes to the duration of the interview. This is a flexible dose, open trial, which means the doctor in charge of the patient will know which medication is being prescribed, and that he will be allowed to adapt the dosage according to what he feels necessary. This research project will allow us to organise a more specialised clinic for the care of first episode manic patients. We will take this opportunity to study carefully the months preceding the appearance of the first episode in order to try to reconstruct the prodrome of bipolar disorders. We will also, in an extension phase of the study, look at the long term outcome (at 6 and 12 months) of a first episode of mania.

DETAILED DESCRIPTION:
This prospective single-centre open trial will compare two groups receiving two different neuroleptics combined with lithium during the first 8 weeks of treatment of a first manic episode. All the patients will also be included in a 6 and 12 months follow-up study and will provide information regarding the prodrome of bipolar illness.

The trial comprises five phases: (1) Recruitment and screening; (2) Baseline assessment; (3) 8 weeks treatment phase; (4) Follow-up.

1. Recruitment and screening The Youth Access Team (YAT) assesses all the patients referred to the Early Psychosis Prevention and Intervention Centre (EPPIC) in order to confirm the diagnosis of first psychotic episode. Patients with a clinical presentation compatible with a diagnosis of first episode mania will be presented to the main investigator or to one of the co-investigators for a screening interview. This interview should take place as soon as possible, and not later than 24 hours after admission. During these 24 hours, the patients will be kept under a treatment of benzodiazepine exclusively.

   Any patient meeting the inclusion criteria (including a Young Mania Rating Scale (YMRS) [37] total scores equal or superior to 20) and none of the exclusion criteria at the screening interview will be informed (as well as his/her family) about the study, and they will receive a Patient Information Sheet. A Consent form will be completed if they agree to take part in the study. Patients under section 12 who are unable to give informed consent: these patients will be asked for consent when they are better. The authorised psychiatrist will be able to give consent to treatment on their behalf until they are well. When they are well and are asked to give consent and they do not give consent, all information gathered on this patient will be removed. If the patient declines to consent to the study, she/he will be offered standard clinical care in EPPIC.
2. Baseline assessment Once informed consent will have been given, and provided the YMRS score 24 hours after admission remains greater than 20, patients will be assessed by a research assistant who will be blind to the treatment during the first 8 weeks of the study.

   ¨ The diagnosis will be based on clinical assessment according to the DSM-IV [38] criteria. It will be confirmed during the first week of the study by results of the Structured Clinical Interview for the DSM-IV, Patient Version (SCID-P) [38].

   ¨ The severity of the illness will be evaluated at baseline with the YMRS, the BPRS, the Clinical Global Impression bipolar version (CGI-BP) [39] and the Global Assessment of Functioning (GAF) [38].

   ¨ The depressive symptoms will be assessed with the 21-item Hamilton Depression Rating Scale (HAMD-21) [40].
   * Substance abuse comorbidity will be assessed during the first week with the PACE Substance Use Questionnaire (PSUQ)
   * Level of functioning will be assessed with the Quality if Life Scale (QLS) [41], the Premorbid Adjustment Scale (PAS) [42] and the Modified Vocational Status Index (MVSI) and the Modified Location Code Index (MLCI) [43] during the first week of treatment. If necessary the participation of relatives will be asked.

   In addition, the subjects will undergo physical examination, including blood test, for safety reasons. Demographic data, vital signs, and details on any concomitant medication and medical history will also be collected.

   ¨ Laboratory tests: Haematology: Haemoglobin, MCH, MCHC, MCV, RBC, WCC, platelets, haematocrit. Biochemistry: Total bilirubin, total protein albumin, AST, ALT, alkaline phosphatase, urea, creatinine, sodium, potassium, prolactin, cholesterol, triglycerides, glucose, thyroid function tests (freeT4 and TSH), prolactine level.
3. 8-week Treatment phase: The Australian Clinical Guidelines for Early Psychosis [44] suggest that first episode patients should ideally be observed during 24 hours before any medication is started. This rule will also be applied in the context of the study. During this period, the medication will be restricted to benzodiazepines except in case of severe agitation. In case of severe agitation neuroleptics will be prescribed, if possible after informed consent and randomisation.

   Patients will thereafter be randomly assigned to one of two groups: olanzapine + lithium, or chlorpromazine + lithium. The raters (research assistant and one psychiatrist in charge of the rating of the side effects) will be blind to the randomisation process and treatment conditions during the first 8 weeks of the trial.

   Each subject will also be allocated to a case manager and a psychiatrist who will be one of the investigators. The psychiatrist in charge of the patient will not be blind to the treatment, and therefore will not do the rating of side effects. A research assistant will conduct all the psychometric assessments across the 12 months of the study and will remain blind to the medication received during the first 8 weeks of the trial. During this eight weeks period, patients will be seen according to clinical needs, and will be met weekly up to week 4 and then on week 6 and 8 for assessment of current levels of psychopathology, the collection of safety data and assessment of compliance. After the first 8 weeks of treatment, the psychiatrist will be free to change the treatment. Neurolpetics will be continued for a minimum of 6 months and lithium for a minimum of 12 months. Lithium serum level will be assessed at day 4 and 7, and then accordingly to the stability of the blood level.
4. Follow-up prospective evaluation:

   In this phase, the aim is to compare the level of side effects under each medication regimen, the subjective well-being and the adherence to the treatment during the first 8 weeks on treatment. Other aims are to assess the efficacy of both treatments, the incidence of depressive symptoms, and the 6 and 12 months outcome.

   ¨ Side-effects will be assessed weekly with the UKU rating scale.
   * Adherence to the medication will be assessed weekly with the Medication Adherence Rating Scale (MARS).
   * Subjective well-being will be assessed with the Drug Attitude Inventory (DAI) and the Subjective Well-Being Under Neuroleptics Scale (SWN) at week 1,4 and 8.
   * The severity of the illness will be prospectively evaluated on a weekly basis until week 4, and then at week 6 and 8, month 6 and month 12 with the YMRS, the BPRS and the CGI-BP.
   * Depressive symptoms will be assessed at the same time lines with the HAMD-21.
   * Substance abuse comorbidity will be reassessed at week 8, month 6 and month 12 with the PSUQ.
   * Change inn the level of functioning will be assessed with the QLS, the PAS and the MVSI and MLCI at month 6 and month 12.
   * Vital signs and weight change will be reassessed at weeks 4 and 8 and at months 6 and 12, or whenever necessary.
   * Laboratory values will be reassessed at week 8, or whenever necessary.

   SUBJECTS TRIAL SAMPLE The aim is to recruit 75 first episode manic patients over a two years period. EPPIC takes care of 60 to 80 first episode manic patients each year and we plan on a recruitment rate of 50%.

   TREATMENT Trial drugs

   Lithium: Lithium will be started at 500mg per day on day one and will be increased to 500 mg bd from day 2. Serum lithium will be assessed on day 4, and the daily dose of lithium will be adapted accordingly. Serum lithium will be assessed again on day 7 and thereafter once or twice a week depending on the previous results. We will aim at keeping the lithium level between 0.5 and 1.0 mEq/l, ideally between 0.8 and 1.0 mEq/l. (Higher levels are not recommended when lithium is prescribed along with antipsychotics [49] Chlorpromazine: Chlorpromazine will be started at 100 mg/day orally and adjusted from day 2 by steps of 50 mg or 100 mg, upwards or downwards. Chlorpromazine will be continued for a minimum of 6 months, and will be interrupted according to the clinical state.

   Olanzapine: Olanzapine will be started at 5mg/day and adjusted by steps of 2.5mg each day according to the clinical picture, upwards or downwards. Olanzapine will be continued for a minimum of 6 months, and will be interrupted according to the clinical state.

   CONCOMITANT MEDICATION All medications (prescribed or over-the-counter medications) that are ongoing at the start of the trial or started during the trial, must be documented in the file.

   The following medications are allowed, under specified circumstances:

   Diazepam: up to 50 mg/day to alleviate severe agitation. Benztropine: up to 4 mg/day, for treatment-emergent extrapyramidal symptoms. Paroxetin: will be prescribed in case of the occurrence of a depressive episode that persists after optimisation of the lithium treatment and interruption of antipsychotics.

   ASSESSMENTS Safety ¨ The frequency of treatment-emergent adverse events (events that first appear or worsen during the study period) will be compared between both groups.

   ¨ The frequency of side effects as rated with the UKU scale will be compared between both groups.

   ¨ Weight gain will be compared between both groups.

   ¨ Frequency of changes in vital signs and laboratory findings will be compared between both groups.

   Subjective well- being

   ¨ Total scores on the DAI and the SWN will be compared between both groups.

   ASSESSMENT OF SECONDARY OBJECTIVES Adherence

   ¨ Degree of adherence to the treatment as scored on the MARS will be compared between both groups.

   Efficacy

   ¨ End point analysis: Mean change in various scales from baseline to week 4 and week 8 will be used to compare the efficacy of the two treatments:

   ¨ Primary efficacy analysis will be assessed by comparing the mean change in theYMRS total score.

   ¨ Secondary efficacy analysis will be assessed by comparing the mean change in CGI-BP total score and in BPRS total score.

   ¨ Response analysis: Response is defined as at least a 50% drop in the total YMRS total score from base line to the 8-weeks end point. Euthymia is defined as a total score on the YMRS of no greater than 12 at end point. The number of patients reaching both of these levels of improvement in both groups will be compared.

   Incidence of depressive episodes ¨ A worsening in the HAMD-21 score of at least 3 points will be used as a definition of a clinically detectable worsening in depressive symptoms.

   Six and 12 months outcome

   Definition of recovery:
   * Syndromic recovery: Eight contiguous weeks [50] during which the patient no longer meets criteria for a manic, mixed, or depressive syndrome. Recovery from each of these syndromes is based on DSM-IV criteria and is operationalised as follows: manic syndrome-no longer meeting the A or B criterion for a manic episode; depressive syndrome-no longer meeting the A criterion for a major depressive episode; mixed syndrome-no longer meeting the A or B criterion for a manic episode and the A criterion for a major depressive episode.
   * Symptomatic recovery: Eight contiguous weeks [50] during which the patient experiences minimal to no psychiatric symptoms, operationalized as follows: Young Mania Rating Scale total score of 5 or less, Hamilton depression scale total score of 10 or less.
   * Relapse: Relapse is defined as the return of symptoms after a remission of less than 8 weeks.
   * Recurrence: Recurrence is defined as return of symptoms after recovery.
   * Functional recovery: Return to premorbid levels of function for at least 8 contiguous weeks [50]. To assess functional recovery, seven of the nine general items from the Premorbid Adjustment Scale are evaluated at the 6 and 12-month follow-up visit for the interval period (excluding ratings of education and abruptness in the change in work associated with the index episode, since these scores can not change). To meet criteria for functional recovery, subjects has to receive Premorbid Adjustment Scale general item interval scores less than or equal to the premorbid rating on five of the seven items and have no interval item score more than 2 points higher than the corresponding premorbid score. Additionally, functional recovery will be considered to be realised if patients return to at least base level on both MLCI and MVSI.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 15 to 29.
* Experiencing a first episode psychosis.
* Meet DSM-IV criteria for bipolar either manic or mixed episode, or schizoaffective disorder manic episode.
* Minimum score of 20 on the YMRS
* Written informed consent to participation.

Exclusion Criteria:

* Patients at immediate risk of committing harm to self or others
* Use of neuroleptics or mood-stabilisers in the two months preceding admission to EPPIC
* Organic mental disease, including mental retardation
* History of clinically significant illness (liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological or metabolic disturbances).
* Clinically relevant biochemical or hematological abnormalities.
* Pregnant or lactating woman
* History of epilepsy
* History of severe drug allergy or hypersensitivity
* Non fluency in English.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2001-10-01; Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Intensity of side effects | 8 weeks
  Intensity of side effects
¨The frequency of treatment-emergent adverse events (events that first appear or worsen during the study period) will be compared between both groups. | 8 weeks
¨The frequency of side effects as rated with the UKU scale will be compared between both groups. | 8 weeks
¨Weight gain will be compared between both groups. | 8 weeks
¨Frequency of changes in vital signs and laboratory findings will be compared between both groups. | 8 weeks
Subjective well being | 8 weeks
¨Total scores on the DAI and the SWN will be compared between both groups. | 8 weeks

SECONDARY OUTCOMES:
Adherence | 8 weeks
¨Degree of adherence to the treatment as scored on the MARS will be compared between both groups. | 8 weeks
Response to treatment | 8 weeks
¨End point analysis: Mean change in various scales from baseline to week 4 and week 8 will be used to compare the efficacy of the two treatments: | 8 weeks
¨Primary efficacy analysis will be assessed by comparing the mean change in theYMRS total score. | 8 weeks
¨Secondary efficacy analysis will be assessed by comparing the mean change in CGI-BP total score and in BPRS total score. | 8 weeks
¨Response analysis: Response is defined as at least a 50% drop in the total YMRS total score from base line to the 8-weeks end point. Euthymia is defined as a total score on the YMRS of no greater than 12 at end point. The number of patients reaching bot | 8 weeks
Incidence of depressive episodes | 8 weeks
¨A worsening in the HAMD-21 score of at least 3 points will be used as a definition of a clinically detectable worsening in depressive symptoms. | 8 weeks
Six and 12 months outcome | 12 months
Definition of recovery: | 12 months
¨Syndromic recovery: Eight contiguous weeks [50] during which the patient no longer meets criteria for a manic, mixed, or depressive syndrome. Recovery from each of these syndromes is based on DSM-IV criteria and is operationalised as follows: manic synd | 12 months
¨Symptomatic recovery: Eight contiguous weeks [50] during which the patient experiences minimal to no psychiatric symptoms, operationalized as follows: Young Mania Rating Scale total score of 5 or less, Hamilton depression scale total score of 10 or les | 12 months
¨Relapse: Relapse is defined as the return of symptoms after a remission of less than 8 weeks. | 12 months
¨Recurrence: Recurrence is defined as return of symptoms after recovery. | 12 months
¨Functional recovery: Return to premorbid levels of function for at least 8 contiguous weeks [50]. To assess functional recovery, seven of the nine general items from the Premorbid Adjustment Scale are evaluated at the 6 and 12-month follow-up visit for | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Conus, Principal Investigator — ORYGEN Youth Health & Department of Psychiatry, The University of Lausanne
Locations (1):
- ORYGEN Youth Health, Parkville, Victoria, Australia